CLINICAL TRIAL: NCT03674216
Title: Prospective Study of Peripherally Inserted Venous Catheters in CF Patients
Brief Title: Study of Peripherally Inserted Venous Catheters in Cystic Fibrosis Patients
Acronym: PICC-CF
Status: Completed | Type: Observational
Sponsor: Jonathan B. Zuckerman (Other)
Collaborators: MaineHealth (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor-Investigator, Jonathan B. Zuckerman, Director, Adult Cystic Fibrosis Program, MaineHealth
Organization: MaineHealth (Other)
Other Study IDs: 1223366
Record Dates: First submitted 2018-09-12; First posted 2018-09-17 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cystic Fibrosis
Keywords: peripherally inserted central venous catheter; midline catheter; thrombosis; blood stream infection
MeSH Terms: conditions — Cystic Fibrosis; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
According to the U.S. CF Foundation Patient Registry, more than 25% of children and 40% of adults were treated with intravenous (IV) antibiotics for flares of lung disease in 2016. Medication for these flares is often delivered through a peripherally inserted central catheter (PICC). Case series have identified important complications of PICCs in CF patients such as blood clots and infection. The frequency of PICC-associated blood clots in CF patients ranges from 2 to 8%. Catheter-related complications may interfere with completion of therapy and lead to repeated procedures and other complex medical treatments. In some cases PICC complications may discourage patients from accepting future courses of IV antibiotics. Therefore, it is very important to identify patient- and device-related factors that are linked with more frequent complications and to figure out ways to reduce these risks. Proposed risk factors fall into several broad categories. First are catheter-related factors; second are patient factors; and third are catheter-management factors. To date, no multicenter trial has carefully studied PICC complications in a large group of adult and pediatric CF patients from the time each catheter is placed to when it is removed. The main purpose of this study is to see whether the investigators can identify important factors in each of the three categories (patient, catheter, and catheter management) that are linked to various complications.

DETAILED DESCRIPTION:
According to data from the U.S. CF Foundation Patient Registry (CFFPR), more than 25% of children and 40% of adults were treated with intravenous (IV) antibiotics for pulmonary exacerbations (PEx) in 2016; this translated to 20,286 care episodes. Case series have identified important complications of PICCs and TIVADs in CF patients such as deep venous thrombosis (DVT) and infection; central venous stenosis; and other types of mechanical dysfunction. The incidence of PICC-associated DVT in CF patients ranges from 2 to 8%. Proposed risk factors in CF patients fall into several broad categories. First are catheter-related factors: larger catheter size, number of catheter lumens, and catheter composition; second are patient factors: lung function, nutritional status, respiratory flora, diabetes status, thrombophilia; and number of previously placed catheters; and third are catheter-management factors: insertion technique and site selection, inpatient versus outpatient care, anticoagulant use, blood sampling practices, and duration of line use. The importance of some of these factors remains controversial, leading some to call for detailed prospective studies of PICC use in specific patient populations. To date, no multicenter trial has prospectively studied PICC and midline complications in adult and pediatric CF patients. The investigators hypothesize that the rate of PICC and midline vascular complications is associated with specific patient level and line level factors as well as with line insertion and management practices. The proposed trial is a multicenter, prospective surveillance study to evaluate (patient level-, catheter level- and catheter management-) risk factors associated with various complications of PICCs and midlines in pediatric and adult CF patients.

ELIGIBILITY:
Inclusion Criteria:

* All ethnic groups
* Females and males
* 6 years of age and above (in order to perform spirometry on all study participants)
* Undergoing treatment for PEx with IV antibiotics via hospital-placed PICC or midline catheter
* Ability to communicate with pertinent staff.
* Ability to understand and willingness to comply with the requirements of the trial (allow repeated assessment of the catheter insertion site, photographs of the site, extremity measurement and face-to face assessment on the day of line removal).
* Ability and willingness to give verbal consent (with the assistance of a parent or guardian, if appropriate) or assent (for pediatric patients)
* Diagnosis of cystic fibrosis consisting of both:

  * sweat sodium or chloride > 60 mEq/L by the pilocarpine iontophoresis method or cystic fibrosis genotype (homozygous for CFTR mutation or compound heterozygous for CFTR mutations)
  * clinical manifestations of cystic fibrosis

Exclusion Criteria:

* Under age 6
* Planned use of a TIVAD or peripheral catheter for IV therapy for the full course of therapy
* History of >10 PICCs prior to study entry
* IV treatment anticipated to extend beyond 21 days at the time of line insertion
* Patient taking anticoagulant medication (other than NSAIDs) at the time of screening
* Inability/unwillingness to provide consent or assent

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric and adult cystic fibrosis patients
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Development of catheter related deep venous thrombosis or catheter occlusion | While the catheter is in place, an average of two weeks
  Occlusion of the catheter requiring removal or symptomatic venous thrombosis in the extremity with the line as indicated by a Constans Clinical Decision Score greater than or equal to 2. The range of the scale goes from -1 to 3 with higher scores representing worse outcome. One point is added to a baseline score of 0 for each of the following: indwelling venous material, localized pain, unilateral pitting edema. One point is subtracted for another diagnosis being at least as plausible as venous thrombosis.

SECONDARY OUTCOMES:
Development of catheter related local phlebitis or superficial thrombophlebitis | While the catheter is in place, an average of two weeks
  Phlebitis as defined by a Visual Infusion Phlebitis (VIP) score greater than or equal to 2. The range of the scale goes from 0 to 5 with higher scores representing worse outcome. The values on the VIP scale are defined as follows: 0-site appears healthy; 1- One of the following: Pain near the IV site or erythema near the IV site; 2- Two of the following: Pain or erythema or swelling near the IV site; 3- All of the following: Pain, erythema, and induration near the IV site; 4- All of the following: Pain, erythema, and palpable venous cord near the IV site; 5- All of the following: Pain, erythema, palpable venous cord and fever >38 degrees centigrade. Thrombophlebitis is defined by phlebitis associated with superficial thrombosis as detected by ultrasound or venogram.
Central line associated blood stream infection (CLABSI) | While the catheter is in place, an average of two weeks
  The study definition for CLABSI follows the Centers for Disease Control guidelines
Number of participants with catheter associated deep venous thrombosis | While the catheter is in place, an average of two weeks
  Deep venous thrombosis as confirmed by ultrasound and/or venogram

OTHER OUTCOMES:
Number of patients with catheter associated hematoma or bleeding | While the catheter is in place, an average of two weeks
  Visible bruising associated with the catheter insertion site, bleeding from the catheter insertion site or incident hemoptysis
Number of patients with catheter associated site pain | While the catheter is in place, an average of two weeks
  Pain in the extremity associated with the catheter
Number of patients with catheter fracture | While the catheter is in place, an average of two weeks
  Catheter fracture
Number of patients with temporary occlusion of the catheter | While the catheter is in place, an average of two weeks
  Temporary occlusion of the catheter cleared by thrombolytic agent
Catheter associated change in arm circumference | While the catheter is in place, an average of two weeks
  Arm circumference in centimeters (cm) measured 5 cm distal to the catheter insertion site
Serum C-reactive protein concentration | While the catheter is in place, an average of two weeks
  Serum measure of inflammatory status with samples taken at the time of catheter insertion and removal
Serum D-dimer concentration | While the catheter is in place, an average of two weeks
  Blood test to assess coagulation status with samples taken at the time of catheter insertion.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Zuckerman, M.D., Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No